CLINICAL TRIAL: NCT01828996
Title: Shocking Therapy for Pelvic Pain: Evaluation of Shock Wave Therapy to Treat Chronic Pelvic Pain in Men
Brief Title: Shocking Therapy for Chronic Pelvic Pain Syndrome
Acronym: CPPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CAN-SW-001
Record Dates: First submitted 2013-03-04; First posted 2013-04-11 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome
Keywords: Chronic pelvic pain syndrome; Chronic prostatitis; Shock wave therapy; Prostate; Pelvic floor; Pain
MeSH Terms: conditions — Prostatitis; Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shock wave therapy (Active Comparator): This group of patient will be treated with the shock wave head in the first 4 sessions then crossover to have the stand-off placebo for another 4 sessions.
  Interventions: Device: Shock wave therapy; Device: Placebo
- Placebo (Placebo Comparator): This group of patient will be treated with the stand-off placebo for the first 4 sessions then crossover to have the shock wave head in the other 4 sessions .
  Interventions: Device: Shock wave therapy; Device: Placebo

INTERVENTIONS:
Device: Shock wave therapy — A total of 3000 pulses will be applied, moving the shock head every 500 pulses to cover the entire prostate and pelvic floor region.
  Other Names: Storz Duolith SD1
Device: Placebo — A total of 3000 pulses will be applied, moving the shock head every 500 pulses to cover the entire prostate and pelvic floor region
  Other Names: Storz Duolith SD1 with stand-off head

SUMMARY:
Chronic prostatitis/chronic pelvic pain syndrome is an extremely common urologic diagnosis and accounts for approximately 2 million outpatient visits to urology practices in the United States alone. Up to 6% of men in Canada recently experienced at least moderate to severe prostatitis-like symptoms with two thirds having symptoms lasting more than one year. There are a myriad of therapies for prostatitis, some of which work on some of the men but none works for all the men. Recently, a number of centres have been using low energy shock waves applied on the skin to target the prostate and the muscles around the prostate. The initial reports showed a significant reduction in the pain experienced by the men with prostatitis. However, this potentially highly promising therapy has not been widely used at least in part due to a lack of properly designed studies to validate this therapy. The investigators plan a randomized control trial using shock wave therapy on men with prostatitis. The goal is to provide some solid evidence that either shock waves are or are not of clinical benefit.

The investigators hypothesize men with chronic prostatitis/ chronic pelvic pain syndrome will have a reduction in pain and improved voiding and sexual function following low power transdermal shock wave therapy to the prostate and surrounding pelvic muscles.

ELIGIBILITY:
Inclusion Criteria:

* Exhibit symptoms of pain typical for prostatitis/CPPS
* Have had the symptoms for at least 3 months
* Have no evidence of infection in the urine or expressed prostatic secretions (the seminal plasma may be substituted if expressed prostatic secretions are not available).
* Have failed at least one therapy for CPPS

Exclusion Criteria:

* Suspected or confirmed to have prostate cancer
* Have a coagulation disorders
* Use anticoagulants
* Have thrombosis
* Have used cortisone therapy up to 6 weeks before first treatment
* Are actively trying to conceive

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in pain | 32 weeks after entering into trial
  Changes in pain is measured by a visual analog scale from question 4 from the NIH- Chronic Prostatitis Symptom Index. The NIH-CPSI is a validated instrument used to measure and follow changes in pain, impact and bother from CPPS.
  We are calculating the changes from the last time point to the first time point (baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Keith Jarvi, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada